CLINICAL TRIAL: NCT04235595
Title: Comparison of the Effects of High-frequency TENS and Connective Tissue Manipulation on the Primary Dysmenorrhea
Brief Title: Comparison of the Effects of TENS and CTM on Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Bakircay University (Other)
Responsible Party: Principal Investigator, Nilay Yürekdeler Şahin, Assistant Professor, Izmir Bakircay University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: primary dysmenorrhea ctm; 2014SBE008 (Other Grant/Funding Number: Pamukkale University Scientific Research Projects)
Record Dates: First submitted 2020-01-13; First posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Primary Dysmenorrhea
Keywords: Primary dysmenorrhea; Connective tissue manipulation (CTM); Transcutaneous electrical nerve stimulation (TENS); Pain
MeSH Terms: conditions — Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Connective Tissue Manipulation (Experimental): The participants were administered CTM by a physiotherapist with 11 years of experience in the application from the point at which their menstrual cycles had ended to the beginning of the next cycle. Another assessment was made immediately after the treatment and this was repeated at the second, third and fourth menstrual cycles. The CTM took an average of 20-30 minutes to complete.
  Interventions: Other: Connective Tissue Manipulation
- Transcutaneous Electrical Nerve Stimulation (Experimental): Following the assessment made in the participants' first menstrual cycle, on the most painful day of their second cycle (1st or 2nd day of the cycle), high-frequency TENS was applied at a frequency of 120 Hertz, at intervals of 100 µsn for 20 minutes. The intensity of the current was increased until the participant felt it.
  Interventions: Other: Transcutaneous Electrical Nerve Stimulation

INTERVENTIONS:
Other: Connective Tissue Manipulation — The application was delivered with the participant in a sitting position, with the entire back and sacral regions left exposed. The treatment was administered to the sacral, lower thoracic and pelvic regions.
  Other Names: CTM
  Arms: Connective Tissue Manipulation
Other: Transcutaneous Electrical Nerve Stimulation — TENS was administered with the participant lying face down with a flat cushion underneath the abdomen. TENS was administered via 2 channels of electrodes placed with the sacral region in the middle. The intensity of the current was increased until the participant felt it.
  Other Names: TENS
  Arms: Transcutaneous Electrical Nerve Stimulation

SUMMARY:
this study was to compare the early and short-term effects of high-frequency transcutaneous electrical nerve stimulation (TENS) versus connective tissue manipulation (CTM) in participants with primary dysmenorrhea. Half of the participants received CTM, while the other half received TENS.

DETAILED DESCRIPTION:
CTM and TENS each relieve dysmenorrhea pain, but they do so by different. The electrotherapy modality that is most commonly used in the treatment of dysmenorrhea is TENS. It has been reported in studies that high-frequency TENS is more effective in reducing pain than either low-frequency TENS or placebo TENS.

A scan of the literature reveals that although there are differing opinions and applications related to the number and duration of CTM, it has been shown that women with primary dysmenorrhea experience reduced pain after CTM,

ELIGIBILITY:
Inclusion Criteria:

* being between the ages of 18-30
* having a diagnosis of primary dysmenorrhea

Exclusion Criteria:

* having used an oral contraceptive in the last 3 months,
* having an active sexual life,
* pregnancy,
* having gone through childbirth,
* having a neurological deficit,
* any kind of systemic condition,
* a diagnosed gynecological condition (pelvic inflammatory diseases, endometriosis, uterus cancers, ovarian cysts, etc.),
* taking psychotherapeutic drugs.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Menstrual cycle
Enrollment: 40 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-03-15 (Actual); Study Completion 2016-08-30 (Actual)

PRIMARY OUTCOMES:
Assessment of Pain Severity | Change from Pain severity at 3 months
  To determine the localization of pain, the participants were asked to point out and mark the place(s) they felt the most pain on a body diagram. The severity of the pain of dysmenorrhea was assessed on a 10-cm Visual Analog Scale (VAS).

SECONDARY OUTCOMES:
Assessment of Sleep Disorders and Fatigue | Change from Sleep Disorders and Fatigue severity at 3 months
  A 10cm VAS was used to assess the severity of sleep disorder and fatigue in the cases of dysmenorrhea.
Assessment of Depressive Symptoms | Change from Beck Depression Inventory score at 3 months
  The Turkish version of the Beck Depression Inventory (BDI) was used in order to identify the risk participants faced in terms of depression and the level of their depressive symptoms. The inventory contains 21 categories, each having 4 choices to mark. The items score between 0-3. The total possible score is 0-63. A score of 0-9 is defined as relating to depressive symptoms at a minimal level, a score of 10-16 to slight depressive symptoms, 17-29 to moderate depressive symptoms, 30-63 to severe depressive symptoms.
Assessment of Anxiety | Change from Beck Anxiety Inventory score at 3 months
  The Turkish version of the Beck Anxiety Inventory (BAI) was used to assess anxiety. This inventory consists of 21 categories, each item being scored on a scale of 0-3. The total possible score on the inventory is 0-63. A score of 0-17 is defined as indicating low, 18-24 as indicating moderate, and a score of 25 and over as indicating a high level of anxiety
Assessment of General Health Status | Change from General Health Questionnaire score at 3 months
  The "General Health Questionnaire" (GHA-28) was used in order to learn the general health status of the participants during their menstrual cycles. The 28-item questionnaire we used in the study assesses the psychological symptoms experienced in the last week. The questionnaire contains four sub-divisions of seven items each. The minimum score on the scale is 0; maximum is 84. Higher scores indicate a state of poor health.

CONTACTS AND LOCATIONS:
Overall Officials: Nesrin Yağcı, Study Director — Pamukkale University

IPD SHARING:
Plan to Share IPD: No